CLINICAL TRIAL: NCT02591706
Title: Clinical and Radiographic Assessment of V3 Implant: A Randomized Controlled Trial
Brief Title: Clinical Assessment of Dental Implant
Acronym: H2015-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Collaborators: MIS Implant Technologies, Ltd (Industry)
Responsible Party: Principal Investigator, Dr. France LAMBERT, Head of Clinic, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H2015-1
Record Dates: First submitted 2015-10-09; First posted 2015-10-29 (Estimated); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Tooth Loss
Keywords: Single missing tooth; Implants; Peri-implant bone remodeling; Bone thickness; Thickness of soft tissue
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dental implant (C1) (Active Comparator): Internal Conical Connection: The C1 has a six-position cone index, except for the C1 narrow platform that has a four-position cone index. The conical connection is 2.00mm in depth, with a 12° cone. As a result of our meticulous manufacturing process a perfect fit between the implant and the abutment is achieved, eliminating micro-movements and minimizing bone resorption.
  Patient will be randomly assigned to one of the two groups after flap opening.
  Interventions: Device: MIS Implants
- Dental implant (V3) (Experimental): The unique triangular shape of the coronal portion of the V3 implant results in less titanium and more bone and soft tissue visible in the esthetic zone, for a restorative-driven approach and easier soft tissue management. The V3 provides doctors with a more advantageous starting point; where greater volume of bone and soft tissue is achieved at the onset of implant placement.
  Patient will be randomly assigned to one of the two groups after flap opening.
  Interventions: Device: MIS Implants

INTERVENTIONS:
Device: MIS Implants — The implantation procedure will be carried out according to a standard surgical protocol, and according the manufacture protocol. Patient will be randomly assigned to one of the two groups after flap opening. The implant stability will be measured using the wench key and recorded in N/cm. The implants will be covered with healing abutments for trans-gingival healing for a period of 4 months. The area will be sutured with thin nylon sutures for a primary passive fit closure. Immediately after the surgery the patient will perform a CBCT of the treated area with a cotton roll on the buccal side in order to be able to evaluate the buccal soft tissue thickness.
  Other Names: MIS Implants Technologies

SUMMARY:
Primary Endpoints : The implant survival and success rate of V3 and C1 implants will be compared. Implant success rate will be evaluated by measuring the peri-implant bone remodeling from baseline to 1 year post insertion.

The hypothesis is those implant survival rates of the test (V3) and control group (C1) are similar and that test V3 implant allows less peri-implant bone loss.

Secondary Endpoints : The thickness of hard tissue in the buccal aspect of the V3 and C1 implants will be compared. The bone thickness will be measured in cone beam computerized tomography (CBCT) on the day of implantation, 4 and at one year after the final restoration.

The hypothesis is that V3 implant allows thicker bone dimension in the cervical area.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have voluntarily signed the informed consent form before any study related action
* Age: 18 with one or more missing teeth in the maxillary area, seeking for implant therapy.
* Men/Women
* In good systemic health (ASA I/ II)
* Present with no contra indication against oral surgical interventions
* Patients required replacement of a single missing tooth. The tooth at the implant site(s) must have been extracted or lost at least 12 weeks before the date of implantation.
* At least 10 mm of bone in the vertical dimension
* At least 6 mm of bone in the bucco-lingual dimension.
* No need for bone augmentation procedure in any of the dimensions
* Full mouth plaque score (FMPI) lower or equal than 25%

Exclusion Criteria:

* Autoimmune disease require medical treatment
* Medical conditions requiring prolonged use of steroids
* Use of Bisphosphonate intravenously or more then
* Infection (local or systemic) - patient with gingivitis or active local infection will undergo a medical treatment prior to his entrance to the study, each individual will be evaluated prior to study procedure for suitability, in case of systemic infection the evaluation will be based on medical anamneses, and if necessary will be referred to relevant medical tests.
* Current pregnancy or breastfeeding women
* Alcoholism or chronically drug abuse
* Immunocompromised patients
* Uncontrolled Diabetes
* Smokers
* Prisoners

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-02-02 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Comparison of implant survival and success rate of V3 and C1 implants | 1 year
  Implant success rate will be evaluated by measuring the peri-implant bone remodeling from baseline to 1 year post insertion. The hypothesis is those implant survival rates of the test (V3) and similar and that test V3 implant allows less peri-implant bone loss.

SECONDARY OUTCOMES:
Comparison of the thickness of hard tissue in the buccal aspect of the V3 and C1 implants | 1 year
  The bone thickness will be measured in cone beam computerized tomography (CBCT) on the day of implantation, 4 and at one year after the final restoration.

OTHER OUTCOMES:
Measurement of aesthetic outcomes based on the pink esthetic score | 1 year
  The mesial papilla, distal papilla, soft tissue level, soft tissue contour, alveolar process deficiency, soft tissue color and texture will be assessed at baseline (crown placement) and at 1 year after the final restoration by using the Pink Esthetics Score (PES).

CONTACTS AND LOCATIONS:
Overall Officials: France LAMBERT, Study Director — University of Liege
Locations (1):
- CHU de Liège - Service de Médecine Dentaire, Liège, Belgium